CLINICAL TRIAL: NCT04762771
Title: Open-label (Unblinded) Randomization to Treatment of Colchicine Plus Current Care Per Institution Treating Physicians vs. Current Care Per Institution Treating Physicians (Control Arm)
Brief Title: Colchicine for the Treatment of Cardiac Injury in Hospitalized Patients With COVID-19 (COLHEART-19)
Acronym: Colheart-19
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recovery Trial showed no convincing evidence that further recruitment would provide conclusive proof of worthwhile benefit for the evaluation of Colchicine in patients with Covid-19.
Sponsor: Baptist Health South Florida (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 152247; NCT04510038 (obsolete NCT alias)
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Results first posted 2022-03-14 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Colchicine; Therapeutics; Standard of Care

STUDY DESIGN:
Intervention Model Description: This is an unblinded randomized study to treat hospitalized covid-19 patients with colchicine plus current care per institution treating physicians vs. current care per institution treating physicians alone (the control arm)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Hospitalized covid-19 patients treated with colchicine plus current care per institution treating physicians.
  Interventions: Drug: Colchicine
- Control (No Intervention): Hospitalized covid-19 patients treated with current standard of care (per institution treating physicians) alone.

INTERVENTIONS:
Drug: Colchicine — Colchicine dosing = 0.6 mg bid x 30 days Decrease dose to 0.3-0.6 mg daily or every other day in setting of gastrointestinal intolerance (nausea, diarrhea, emesis, abdominal discomfort) Decrease dose to 0.6 mg daily in the setting of weak or moderate CYP3A4 inhibitor Decrease dose to 0.3 mg daily in the setting of strong CYP3A4, P-glycoprotein inhibitors, or protease inhibitors Decrease dose to 0.3 mg daily in the setting of chronic kidney disease (CKD) stage ≥ 4 (CrCl ≤ 30 ml/min) or liver failure (aspartate aminotransferase /alanine aminotransferase > 3x normal).
  Decrease dose to 0.6 mg every 14 days in patients with end stage renal disease (ESRD) or requiring dialysis Route of Administration: oral
  Other Names: Treatment with Colchicine plus standard of care in hospitalized patients with Covid-19
  Arms: Active

SUMMARY:
This is an open-label unblinded, randomized study to treat hospitalized covid-19 patients with colchicine plus current care (per institution treating physicians) vs. current care per institution treating physicians alone (the control arm)

DETAILED DESCRIPTION:
We aim to determine if Colchicine improves short-term outcomes in hospitalized coronavirus disease-19 (COVID-19) patients with cardiac manifestations of disease.

Myocardial injury has been described in up to 30% of COVID-19 infected patients, and portends a poor prognosis with currently no known treatment. Colchicine is a widely available, well-established, inexpensive, oral anti-inflammatory agent that has been FDA approved for the treatment of inflammatory disorders including gout and familial Mediterranean Fever. Trials have also shown its benefit to prevent post-cardiotomy syndrome, to treat acute and recurrent pericarditis, and reduce cardiovascular events after myocardial infarction. We extrapolate based on these indications and studies that colchicine may also help improve outcomes in hospitalized COVID-19 patients with evidence of cardiac injury.

This is an unblinded randomized study to treat hospitalized covid-19 patients with colchicine plus current care per institution treating physicians vs. current care per institution treating physicians alone (the control arm)

ELIGIBILITY:
Inclusion Criteria:

* Men and Women ≥ 18 years of age
* Covid-19 Positive
* Hospitalized patients able to provide informed consent
* Cardiac injury (as evidenced by any of the following)

  1. Elevated troponin level
  2. Elevated BNP level
  3. New ischemic or arrhythmogenic ECG/telemetry changes
  4. New decrease in Left Ventricular Ejection Fraction (LVEF) or new pericardial effusion on echocardiogram

Exclusion Criteria:

* Pregnancy, breastfeeding mothers, and women of childbearing age who are unable to use adequate contraception, which includes:

  1. Intrauterine devices (IUD), contraceptive implants, or tubal sterilization
  2. Hormone method with a barrier method
  3. Two barrier methods
  4. If a partner's vasectomy is the chosen method of contraception, a hormone or barrier method must also be used in conjunction
* History of severe hematologic or neuromuscular disorder
* Co-administration of Cytochrome P450 3A4 (CYPA3A4) and P-glycoprotein transport inhibitor
* Severe renal impairment with concomitant hepatic impairment
* Concurrent use of colchicine and strong or P-glycoprotein inhibitor with renal or hepatic impairment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2021-05-12 (Actual); Study Completion 2021-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Chaparro, MD, Principal Investigator — Baptist Health South Florida; Raul E Herrera, MD, Study Director — Baptist Health South Florida
Locations (1):
- Baptist Hospital of Miami, Miami, Florida, United States

REFERENCES:
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The rapid decline in COVID patients and other competing trials did not allowed enrollment of additional subjects. Given the small sample size, the study was terminated.
Pre-assignment Details: Patients who test positive for COVID-19, sign informed consent and have any of the study specific manifestations of cardiac injury were randomized 1:1 .
Groups:
- Control - Standard of Care Alone: Hospitalized covid-19 patients treated with current standard of care (per institution treating physicians) alone.
- Active - Colchicine Plus Standard of Care: Hospitalized covid-19 patients treated with colchicine plus current care per institution treating physicians.
  Colchicine: Colchicine dosing = 0.6 mg bid x 30 days Decrease dose to 0.3-0.6 mg daily or every other day in setting of gastrointestinal intolerance (nausea, diarrhea, emesis, abdominal discomfort) Decrease dose to 0.6 mg daily in the setting of weak or moderate CYP3A4 inhibitor Decrease dose to 0.3 mg daily in the setting of strong CYP3A4, P-glycoprotein inhibitors, or protease inhibitors Decrease dose to 0.3 mg daily in the setting of chronic kidney disease (CKD) stage ≥ 4 (CrCl ≤ 30 ml/min) or liver failure (aspartate aminotransferase /alanine aminotransferase > 3x normal).
  Decrease dose to 0.6 mg every 14 days in patients with end stage renal disease (ESRD) or requiring dialysis Route of Administration: oral
Period: Overall Study
Arm/Group | Control - Standard of Care Alone | Active - Colchicine Plus Standard of Care
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active: Hospitalized covid-19 patients treated with colchicine plus current care per institution treating physicians.
  Colchicine: Colchicine dosing = 0.6 mg bid x 30 days Decrease dose to 0.3-0.6 mg daily or every other day in setting of gastrointestinal intolerance (nausea, diarrhea, emesis, abdominal discomfort) Decrease dose to 0.6 mg daily in the setting of weak or moderate CYP3A4 inhibitor Decrease dose to 0.3 mg daily in the setting of strong CYP3A4, P-glycoprotein inhibitors, or protease inhibitors Decrease dose to 0.3 mg daily in the setting of chronic kidney disease (CKD) stage ≥ 4 (CrCl ≤ 30 ml/min) or liver failure (aspartate aminotransferase /alanine aminotransferase > 3x normal).
  Decrease dose to 0.6 mg every 14 days in patients with end stage renal disease (ESRD) or requiring dialysis Route of Administration: oral
- Total: Total of all reporting groups
Arm/Group | Active | Control | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 0 | 1 | 1
  Non-Hispanic | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mortality
Description: Composite of all-cause mortality
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Control
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

2. Primary Outcome: Mechanical Ventilation
Description: Need for mechanical ventilation
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Control
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

3. Primary Outcome: Mechanical Circulatory Support
Description: Need for mechanical circulatory support
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Control
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

4. Secondary Outcome: Time (Days) to the Primary End Point
Description: Number of days from start of therapy to either mortality or need for Mechanical Ventilation or Mechanical Circulatory Support
Time Frame: 90 days
Measure: Number; unit: days
Arm/Group | Active | Control
Number analyzed (Participants) | 1 | 1
days | 0 | 0

5. Secondary Outcome: Peak and Delta (Change From Baseline) Troponin Level
Description: Change from baseline to the time when Troponin levels peak during the hospitalization
Time Frame: baseline and 90 days
Measure: Number; unit: ng/ml
Arm/Group | Active | Control
Number analyzed (Participants) | 1 | 1
ng/ml
  Baseline (Peak) | 0.16 | 0.02
  Delta | -0.07 | 0

6. Secondary Outcome: Baseline Brain Natriuretic Peptide (BNP) Level
Description: Documenting baseline Brain Natriuretic Peptide (BNP) at the time of hospitalization
Time Frame: baseline
Measure: Number; unit: pg/ml
Arm/Group | Active | Control
Number analyzed (Participants) | 1 | 1
pg/ml | 27 | 205

7. Secondary Outcome: Inflammatory Biomarkers
Description: Baseline and delta (change from baseline) of C-Reactive Protein
Time Frame: baseline and 90 days
Measure: Number; unit: mg/l
Arm/Group | Active | Control
Number analyzed (Participants) | 1 | 1
mg/l
  Baseline | 34.2 | 3.0
  Delta | 19.1 | -0.1

8. Secondary Outcome: Hospital Length of Stay
Description: Duration of Hospitalization on each arm
Time Frame: 90 days
Measure: Number; unit: days
Arm/Group | Active | Control
Number analyzed (Participants) | 1 | 1
days | 5 | 14

9. Secondary Outcome: Need for Re-hospitalization
Description: 90-day re-hospitalization rate
Time Frame: 90 days
Measure: Number; unit: times hospitalized
Arm/Group | Active | Control
Number analyzed (Participants) | 1 | 1
times hospitalized | 1 | 2

10. Secondary Outcome: Change in Inflammatory Biomarkers
Description: Baseline and delta (change from baseline) of D-Dimer
Time Frame: baseline and 90 days
Measure: Number; unit: mcg/ml
Arm/Group | Active | Control
Number analyzed (Participants) | 1 | 1
mcg/ml
  Baseline | 0.46 | 0.27
  Delta | 19 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from baseline through the 90 day follow-up period.
Arm/Group | Active | Control
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active (N=1) | Control (N=1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Hospitalization due to COVID-19

LIMITATIONS AND CAVEATS:
The rapid decline in COVID patients and other competing trials did not allowed enrollment of additional subjects. Given the small sample size, the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT04762771/Prot_SAP_001.pdf